CLINICAL TRIAL: NCT05414487
Title: Exploring the Effects of B Cell Depletion With Ofatumumab on Immune Cells and Meningeal Lymphatic Drainage in Patients With Demyelinating Diseases - a Prospective Observational Study
Brief Title: Effects of Ofatumumab Treatment on Immune Cells and Meningeal Lymphatic Drainage in Patients With Demyelinating Diseases
Acronym: OMNISCIENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Chao Zhang, Professor, Tianjin Medical University General Hospital
Other Study IDs: COMB157GCN02T
Record Dates: First submitted 2022-06-06; First posted 2022-06-10 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder; Demyelinating Diseases of the Central Nervous System
Keywords: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder; Demyelinating Diseases; Ofatumumab; Meningeal Lymphatic Drainage
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Demyelinating Diseases | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ofatumumab: 17 RMS patients and 17 NMOSD patients prescribed with Ofatumumab will be enrolled after informed consent.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — There is no treatment allocation. Patients with MS or NMOSD administered Ofatumumab by prescription will be enrolled. Participants will receive 20mg ofatumumab (20 mg/0.4 ml) by subcutaneous injection. Ofatumumab is administrated at baseline, Day 7, Day 14 and monthly thereafter until the end of the study.

SUMMARY:
This is an uncontrolled, prospective, observational cohort study to assess the function of meningeal lymphatic drainage and dynamics of immune cells in patients with relapsing multiple sclerosis (RMS) or Neuromyelitis optica spectrum disorder (NMOSD) after receiving ofatumumab treatment over an observational period of 12 months.

DETAILED DESCRIPTION:
This is an uncontrolled, prospective, observational cohort study in patients with RMS or NMOSD who will receive ofatumumab treatment over an observational period of 12 month. Ofatumumab was administrated 20mg by subcutaneous injection on Days 1, 7 and 14 for initial loading, followed by monthly infusion up to 12 months. Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) will be performed to assess meningeal lymphatic flow in participants before and after ofatumumab treatment.The change of immune cell landscape in RMS or NMOSD patients after receiving ofatumumab treatment will be monitored by mass cytometry (CyTOF). Assessments also include clinical assessments( clinical relapse rate and EDSS score) and MRI assessments (T2 lesion load, T1 gadolinium enhancing lesion number).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. RRMS subtype according to 2017 McDonald diagnostic criteria
3. Diagnosis of NMOSD according to the 2015 International Panel diagnostic criteria for NMOSD with AQP4-IgG
4. Newly diagnosed with MS/NMOSD and initiating ofatumumab treatment within the next 3 months

Exclusion Criteria:

1. Hypersensitivity to trial medications
2. History of life-threatening reaction to Ofatumumab
3. Acute or uncontrolled chronic medical condition
4. Have been treated with medications as specified or within timeframes specified (e.g. corticosteroids, rituximab, ocrelizumab, alemtuzumab, natalizumab, cyclophosphamide, claridbine, etc.)
5. Impaired hearing
6. Claustrophobia
7. 300 lbs of greater (weight limit of MRI table)
8. Pregnancy or breastfeeding
9. Sensitivity to imaging agents
10. Contraindications to MRI
11. Use of benzodiazepines, topiramate, doxycycline, mynocicline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. 17 patients with relapsing remitting multiple sclerosis（RRMS）received ofatumumab treatment were enrolled.
  2. 17 patients with NMOSD received ofatumumab treatment were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Time to Peak (TTP) of the meningeal lymphatic vessels in superior sagittal sinus (mLVs-SSS) to the end of study. | Baseline, Up To 12months (End of Study)
  The image of mLVs-SSS in participants will be detected by Dynamic contrast-enhanced MRI (DCE-MRI) before and after ofatumumab treatment.MRI images would be analyzed by three radiologists independently, and each of them is blinded to the patients' information. The obtained DCE-MRI data are interpreted semi-quantitatively to generate TTP.

SECONDARY OUTCOMES:
Immune cells landscape over time | Baseline, month 3, month 6, month 12
  The dynamics of immune cells in participants will be detected by mass cytometry (CyTOF) before and after ofatumumab treatment.
Adjudicated On-trial Annualized Relapse Rate (ARR) | Baseline, Up To 12months (End of Study)
  The adjudicated On-trial ARR was computed as the total number of relapses divided by the total number of patient years in the study period. A central independent committee was used to adjudicate all On-trial Relapses as determined by the treating physician. Results reported as adjusted adjudicated On-trial ARR based on a Poisson regression adjusted for randomization strata and historical ARR in 24 months prior to Screening.
Percentage of Participants With Worsening in Expanded Disability Severity Scale (EDSS) Score From Baseline to the end of study | Baseline, Up To 12months (End of Study)
  Disease-related disability was measured by the EDSS before and after ofatumumab treatment. The EDSS was an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments.
Percentage of participants with new lesions by MRI assessments from baseline to the end of study | Baseline, Up To 12months (End of Study)
  Magnetic Resonance Imaging (MRI) will be used to measure presence of increase in number of gadolinium enhancing lesions and T2 lesion load. Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center and evaluated for quality, completeness and adherence to the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Zhang, M.D., Ph.D., Principal Investigator — Department of Neurology, Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bar-Or A, Li R. Cellular immunology of relapsing multiple sclerosis: interactions, checks, and balances. Lancet Neurol. 2021 Jun;20(6):470-483. doi: 10.1016/S1474-4422(21)00063-6. Epub 2021 Apr 27. PMID 33930317
- [Background] Couloume L, Ferrant J, Le Gallou S, Mandon M, Jean R, Bescher N, Zephir H, Edan G, Thouvenot E, Ruet A, Debouverie M, Tarte K, Ame P, Roussel M, Michel L. Mass Cytometry Identifies Expansion of T-bet+ B Cells and CD206+ Monocytes in Early Multiple Sclerosis. Front Immunol. 2021 May 4;12:653577. doi: 10.3389/fimmu.2021.653577. eCollection 2021. PMID 34017332
- [Background] Hershenhouse KS, Shauly O, Gould DJ, Patel KM. Meningeal Lymphatics: A Review and Future Directions From a Clinical Perspective. Neurosci Insights. 2019 Dec 31;14:1179069519889027. doi: 10.1177/1179069519889027. eCollection 2019. PMID 32363346
- [Background] Migotto MA, Mardon K, Orian J, Weckbecker G, Kneuer R, Bhalla R, Reutens DC. Efficient Distribution of a Novel Zirconium-89 Labeled Anti-cd20 Antibody Following Subcutaneous and Intravenous Administration in Control and Experimental Autoimmune Encephalomyelitis-Variant Mice. Front Immunol. 2019 Oct 18;10:2437. doi: 10.3389/fimmu.2019.02437. eCollection 2019. PMID 31681317
- [Background] Louveau A, Herz J, Alme MN, Salvador AF, Dong MQ, Viar KE, Herod SG, Knopp J, Setliff JC, Lupi AL, Da Mesquita S, Frost EL, Gaultier A, Harris TH, Cao R, Hu S, Lukens JR, Smirnov I, Overall CC, Oliver G, Kipnis J. CNS lymphatic drainage and neuroinflammation are regulated by meningeal lymphatic vasculature. Nat Neurosci. 2018 Oct;21(10):1380-1391. doi: 10.1038/s41593-018-0227-9. Epub 2018 Sep 17. PMID 30224810
- [Background] Wang X, Tian H, Liu H, Liang D, Qin C, Zhu Q, Meng L, Fu Y, Xu S, Zhai Y, Ding X, Wang X. Impaired Meningeal Lymphatic Flow in NMOSD Patients With Acute Attack. Front Immunol. 2021 Jun 14;12:692051. doi: 10.3389/fimmu.2021.692051. eCollection 2021. PMID 34194440
- [Background] Zhang C, Zhang TX, Liu Y, Jia D, Zeng P, Du C, Yuan M, Liu Q, Wang Y, Shi FD. B-Cell Compartmental Features and Molecular Basis for Therapy in Autoimmune Disease. Neurol Neuroimmunol Neuroinflamm. 2021 Aug 31;8(6):e1070. doi: 10.1212/NXI.0000000000001070. Print 2021 Nov. PMID 34465614
- [Background] Leipold MD, Maecker HT. Mass cytometry: protocol for daily tuning and running cell samples on a CyTOF mass cytometer. J Vis Exp. 2012 Nov 2;(69):e4398. doi: 10.3791/4398. PMID 23149654
- [Background] Thrash EM, Kleinsteuber K, Hathaway ES, Nazzaro M, Haas E, Hodi FS, Severgnini M. High-Throughput Mass Cytometry Staining for Immunophenotyping Clinical Samples. STAR Protoc. 2020 Jun 30;1(2):100055. doi: 10.1016/j.xpro.2020.100055. eCollection 2020 Sep 18. PMID 33111099
- [Background] Ding XB, Wang XX, Xia DH, Liu H, Tian HY, Fu Y, Chen YK, Qin C, Wang JQ, Xiang Z, Zhang ZX, Cao QC, Wang W, Li JY, Wu E, Tang BS, Ma MM, Teng JF, Wang XJ. Impaired meningeal lymphatic drainage in patients with idiopathic Parkinson's disease. Nat Med. 2021 Mar;27(3):411-418. doi: 10.1038/s41591-020-01198-1. Epub 2021 Jan 18. PMID 33462448
- [Derived] Yang S, Zhang TX, Liu J, Liu Z, Zhu L, Li YY, Feng B, Fan M, Shi FD, Zhang C. Reconstitution of CXCR3+ CCR6+ Th17.1-Like T Cells in Response to Ofatumumab Therapy in Patients With Multiple Sclerosis. Ann Clin Transl Neurol. 2025 May;12(5):1043-1053. doi: 10.1002/acn3.70042. Epub 2025 Mar 31. PMID 40164501